CLINICAL TRIAL: NCT02397031
Title: Randomized, Active-controlled, Clinical Trial Comparing Effects of Mindfulness and Interpersonal Effectiveness Skills in Borderline Personality Disorder
Brief Title: Mindfulness and Interpersonal Effectiveness Skills in Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Juan Carlos Pascual, Psychiatrist, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-MOD-2011-147
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; mindfulness
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness (Experimental): As proposed in dialectical behavioral therapy, mindfulness training consist of a set of behavioral skills that aim at improving patient's attentional control and emotional regulation.
  Interventions: Behavioral: Mindfulness
- Interpersonal effectiveness (Active Comparator): Interpersonal effectiveness skills are focused on improving interpersonal relationships and enhancing patient's ability to display social effective behavior.
  Interventions: Behavioral: interpersonal effectiveness

INTERVENTIONS:
Behavioral: Mindfulness — weekly psychotherapy sessions for 10 weeks (120 min each)
  Arms: Mindfulness
Behavioral: interpersonal effectiveness — weekly psychotherapy sessions for 10 weeks (120 min each)
  Arms: Interpersonal effectiveness

SUMMARY:
The purpose of the study was to determine whether mindfulness training could be more effective than another active intervention in reducing borderline personality disorder (BPD) symptoms. The main hypothesis was that patients allocated to the mindfulness group would show a greater improvement on global BPD symptomatology. As a second objective, we explored some of the possible underlying mechanisms of both active treatments. For that purpose, changes in decentering, mindfulness facets and cognitive processing of social interactions were also evaluated.

DETAILED DESCRIPTION:
The present study aimed at evaluating the efficacy of mindfulness skills (M) versus interpersonal effectiveness skills (IE) on borderline symptoms. For that purpose, a randomized, active-controlled clinical trial was designed. 64 participants with borderline personality disorder (BPD) diagnosis were allocated to mindfulness (n=32) or interpersonal effectiveness skills (n=32). Both interventions were delivered over a 10-week period. The borderline symptom list (BSL-23) was elected as the primary outcome measure. Mindfulness related capacities, decentering and cognitive processing of social interactions were also evaluated with the Five Facet Mindfulness Questionnaire (FFMQ), the Experiences Questionnaire (EQ) and the Multidimensional Scale of Social Expression (EMES-C), respectively. Assessments were conducted pre and post interventions.

ELIGIBILITY:
Inclusion criteria:

* Ages between 18 and 45 years
* BPD criteria according to two diagnostic interviews (SCID-II and DIB-R)

Exclusion Criteria:

* Lifetime diagnosis of schizophrenia, drug-induced psychosis, organic brain syndrome, bipolar disorder or mental retardation
* Participating in any sort of psychotherapy during the study or having participated in dialectical behavioral therapy groups in the past

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
change from baseline in borderline symptoms after a 10 week intervention | 10 weeks
  participants were assessed pre and post interventions

SECONDARY OUTCOMES:
change from baseline in decentering after a 10 week intervention | 10 weeks
  participants were assessed pre and post interventions
change from baseline in mindfulness facets after a 10 week intervention | 10 weeks
  participants were assessed pre and post interventions
change from baseline in social interactions after a 10 week intervention | 10 weeks
  participants were assessed pre and post interventions

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Pascual, PhD, Principal Investigator — Servei de Psiquitria. Hospital de la Santa Creu i Sant Pau

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Soler J, Elices M, Pascual JC, Martin-Blanco A, Feliu-Soler A, Carmona C, Portella MJ. Effects of mindfulness training on different components of impulsivity in borderline personality disorder: results from a pilot randomized study. Borderline Personal Disord Emot Dysregul. 2016 Jan 11;3:1. doi: 10.1186/s40479-015-0035-8. eCollection 2016. PMID 26759718